CLINICAL TRIAL: NCT06448702
Title: Evaluation of Efficacy and Safety of Enhanced External Counter-pulsation on Patients With Atopic Dermatitis and Inflammatory Skin Disease Requiring Wet Wrap Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HKWC-2024-295
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis; Inflammatory Skin Disease
Keywords: atopic dermatitis; wet wrap therapy; Enhanced External Counter-pulsation
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wet wrap therapy (WWT) (Active Comparator): WWT with mometasone propionate ointment: paraffin soft white 1: 10: once daily (45 minutes ± 15 minutes) x 3 times ±1 time (day 1, day 3, day 5 or any 3 days over 7days, subject to patient self-assessment).
  For those who do not achieve EASI50 (50% reduction of baseline EASI) or EASI<10 on Day 7, they will be asked to enroll to another arm (EECP arm), and have a follow-up visit on Day 14 and 4 weeks post last treatment.
  Interventions: Procedure: wet wrap therapy; Device: External compression counter-pulsation (EECP)
- EECP therapy (Active Comparator): EECP therapy once daily x 3 times ±1: Day 1, Day 3, Day 5 (or any 3 days over 7 days).
  For those who do not achieve EASI50 or EASI total score < 10 on day 7,(or BSA>5%) they will be asked to continue for one more cycle (i.e. 3 more EECP sessions over the next 7 days), and will be followed up on Day 14 and at week 4 post-treatment.
  Interventions: Device: External compression counter-pulsation (EECP)

INTERVENTIONS:
Procedure: wet wrap therapy — Steps for wet wrap therapy After bath/shower with emollients, pat to remove excess water on body and apply the emollient and/ or steroid cream liberally on the affected area to enhance water absorption and seal in moisture Put wet wrap garment in lukewarm water, squeeze water out of the wet wrap garment, take them out without dribbling of water and then apply on the affected area Put on another layer of dry garments/ warm clothing to cover the wet wrap garments and wear usual clothing as needed Check regularly and keep the wet wrap garments underneath damp with water sprayer or wet towel if necessary Patient is suggested to apply emollients frequently throughout the day to maintain the effect
  Arms: wet wrap therapy (WWT)
Device: External compression counter-pulsation (EECP) — External compression counter-pulsation (EECP) is a compression/decompression non-invasive device (Stendo Pulsewave ® V3 CE certificate class IIa) used for lower part of the body (legs, thighs and buttock/hips) to reproduce and stimulate the natural physiological pulsations and the physical shear stress force.

SUMMARY:
Patients with atopic dermatitis (AD) and erythematous skin disease are often treated with topical treatment containing corticosteroids. However, long term use of topical corticosteroid is well known for its potential side-effects such as skin atrophy, hirsutism, dyspigmentation, telangiectasia, and possible skin infection and iatrogenic adrenal insufficiency. Fear about medication side effects would cause lack of adherence to treatment regiments and thus patients would seek for alternative therapies, and a long term safer and affordable treatment modality is required to fill this therapeutic gap.

Enhanced external counter-pulsation (EECP) therapy is a non-invasive method to improve perfusion of vital organs and reduces hypercholesterolemia-induced endothelial damage. It also helped to increase cerebral blood circulation in patients with ischemic stroke and improved neurological recovery.

This study aim to evaluate the efficacy and safety of patients with atopic dermatitis and erythematous/ inflammatory skin diseases to receive EECP therapy combined treatment compared to wet wrap therapy alone.

DETAILED DESCRIPTION:
Patients with atopic dermatitis (AD) and erythematous skin disease are often treated with topical treatment containing corticosteroids1 -4. However, long term use of topical corticosteroid is well known for its potential side-effects such as skin atrophy, hirsutism, dyspigmentation, telangiectasia, and possible skin infection and iatrogenic adrenal insufficiency3, 4. Other topical and systemic treatment has been suggested to control atopic dermatitis and other inflammatory skin disorders such as calcineurin inhibitors, phototherapy and immunosuppressants4. Patients may need to use in repeated courses according to the skin condition, and may experience flare if treatment is discontinued and they have to continue with potential side-effects such as organ impairment and immunocompromised state secondary to systemic immunosuppressants. In our practice, wet wrap therapy (WWT) is one of the treatment options for patients with moderate-to-severe AD and some other erythematous/ inflammatory skin disease and WWT has a relatively fast onset in disease -control especially during a flare. New biologics or small molecule inhibitors such as anti-Interleukin 4 or 13 and Januse kinase (JAK) inhibitor are new treatment modality but the cost is high and may not be affordable to all patients1, 5. The fear of potential side effects of local/ systemic treatment may result in poor compliance, and prompting patients to explore alternative therapies. Therefore, a long-term safe and affordable treatment modality is required to fill this therapeutic gap5.

Enhanced external counter-pulsation (EECP) therapy is a non-invasive method to improve perfusion of vital organs and has been proved to reduce hypercholesterolemia-induced endothelial damage6. It operates by applying ECG-triggered pressure to the lower extremities during diastole by means of air-filled cuffs, thus, augmenting diastolic blood flow and reducing systolic afterload. These, in turns, increases blood flow to the heart, brain and kidneys. It has been proved to be effective in increasing the sheer stress of blood vessel and decreasing risk of hypercholesterolemia-induced atherosclerosis by increasing the nitrite oxidase level in blood circulation, which has antiatherogenic, antithrombotic and anti-inflammatory effects6. In human subjects, EECP has also been proved to be effective in improving blood glucose level in patients with diabetes mellitus7, 8. It also helped to increase cerebral blood circulation in patients with ischemic stroke and improved neurological recovery9.

However, there is no pervious study of EECP in patients with atopic dermatitis and erythematous /inflammatory skin diseases. There are various studies showing that vascular inflammation in moderate -to -severe AD patients is associated with enhanced Th2 response10-12. In addition, morphology of blood vessels was abnormal in patients with AD11 and AD patients has higher risks of cardiovascular comorbidities due to the chronic skin inflammation12-13. Therefore, using EECP may be an effective adjunct therapy to AD patients to improve circulation and reduce the inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 to 65 years old present with atopic dermatitis or erythematous / inflammatory skin diseases attending Queen Mary Hospital dermatology clinics requiring wet-wrap therapy (WWT) will be screened for recruitment by attending dermatologist(s)
2. Patients with AD having EASI>10 or erythematous/inflammatory skin disorder BSA>5%
3. Body weight ≥ 40kg at screening and baseline visit
4. Body height ≥ 150cm at screening and baseline visit
5. Patients fulfilling both inclusion and exclusion criteria (stated below) will be recruited for this study after an informed consent has been given.

Exclusion Criteria:

1. Patients who refuse to give consent
2. Females of childbearing potential who are pregnant or during breastfeeding period
3. Patients have newly started systemic corticosteroid, immunosuppressants or biologics within 6 week of Baseline (Day 0)
4. Patients who have unstable AD or inflammatory skin disease, active infection or contagious skin symptoms within 2 weeks before day 1 pre-enrolment
5. Patients who have uncontrolled hypertension, ischemic heart disease or any uncontrolled medical illness
6. Patients who have metallic implants or previous fracture of lower limbs, history of deep vein thrombosis or lower limb varicosity (such as varicose vein), untreated malignancy
7. Patients who cannot tolerate pressure-cuffing, placing in a horizontal position without arching the back or non-compliance to treatment
8. Patients who are taking anticoagulants/ antiplatelet or having bleeding tendency
9. Patients who are having undergone recent major surgery
10. Patients who have a history of phlebitis with acute thrombotic risk
11. Patient who are suffering from an acute disease during the screening period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
EECP therapy treatment should have more superior result compared to those receiving WWT alone | Day 7
  Patients with atopic dermatitis +/- erythematous/inflammatory skin disorders receiving EECP therapy treatment should have more mean reduction of total Eczema Area and Severity Index (EASI) score from baseline to Day 7 compared to those receiving WWT alone.
  EASI score ranges from 0-72, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
achieve EASI 25%/ 50%/ 75% reduction on Day 7 | Day 7
  1. Percentage of participants who achieve EASI 25%/ 50%/ 75% reduction on Day 7 (after the first week of treatment)
second week of treatment and achieve EASI 25%/ 50%/ 75% reduction on Day 14 | Day 14
  2. Percentage of subjects who receive the second week of treatment and achieve EASI 25%/ 50%/ 75% reduction on Day 14 after the second week of treatment
at least 2 points decrease of itch score/sleep score decrease from Baseline visit | Day 7 and or Day 14
  3. Percentage of participants who have at least 2 points decrease of itch score/sleep score decrease from Baseline visit to Day 7 and or day 14 and 4 weeks- post treatment
least 2-point vIGA/ PGA decrease from baseline | Day 14
  4. Percentage of participants who receive the second week of treatment and achieve at least 2-point vIGA/ PGA decrease from baseline 50% reduction comparing to Day 14

IPD SHARING:
Plan to Share IPD: No